CLINICAL TRIAL: NCT00316277
Title: A Two-Phase Randomized Controlled Clinical Trial of Buprenorphine/Naloxone Treatment Plus Standard Medical Management or Enhanced Medical Management for Opioid Analgesic Dependence
Brief Title: Prescription Opioid Addiction Treatment Study (POATS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mclean Hospital (Other)
Collaborators: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Roger D. Weiss, Chief Divsion of Alcohol and Drug Abuse; Professor of Psychiatry, Mclean Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIDA-CTN-0030
Record Dates: First submitted 2006-04-18; First posted 2006-04-20 (Estimated); Results first posted 2012-07-27 (Estimated); Last update posted 2013-02-06 (Estimated); Status verified 2013-02

CONDITIONS: Opiate Dependence; Substance-related Disorders; Opioid-related Disorders
Keywords: Opiate Analgesic Dependence
MeSH Terms: conditions — Opioid-Related Disorders; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Buprenorphine/Nx with EMM (Experimental)
  Interventions: Behavioral: Enhanced Medical Management (EMM) of Prescription Opiate Abuse
- Buprenorphine/Nx with SMM (Active Comparator)
  Interventions: Behavioral: Standard Medical Management (SMM) of Prescription Opiate Abuse

INTERVENTIONS:
Behavioral: Standard Medical Management (SMM) of Prescription Opiate Abuse — Standard Medical Management in Phase 1 will consist of one hour-long initial visit; one individual 15-20 minute visit later in Week 1; one individual 15-20 minute visit per week through the end of Week 4; one 15-20 minute SMM visit at Week 6 and at Week 8. And in Phase 2, one 30-60 minute initial visit; one 15-20 minute follow-up visit later in Week 1; one individual session (15-20 minutes) per week through Week 12. In addition, participants in Phase 1 will receive BUP/NX at between 8 to 32mg/day; tapering to zero between weeks three and four. Those referred to Phase 2 will receive up to 32 mg/day for three months tapering to zero during month four.
  Arms: Buprenorphine/Nx with SMM
Behavioral: Enhanced Medical Management (EMM) of Prescription Opiate Abuse — Enhanced Medical Management in Phase 1 will consist of SMM plus two individual sessions with a counselor per week (45 minutes each) through Weeks 1-4, and one 45-minute counseling visit at Week 6 and at Week 8. And in Phase 2, EMM will consist of the SMM plus two individual sessions with a counselor per week (45 minutes each) during Weeks 1-6 and one individual session with a counselor per week (45 minutes each) during Weeks 7-12. In addition, participants in Phase 1 will receive BUP/NX at between 8 to 32mg/day; tapering to zero between weeks three and four. Those referred to Phase 2 will receive up to 32 mg/day for three months tapering to zero during month four.
  Arms: Buprenorphine/Nx with EMM

SUMMARY:
The purpose of this study is to determine whether treatment outcome for subjects dependent on prescription opioid analgesics can be improved by adding individual drug counseling to the prescription of buprenorphine/naloxone with standard medical management. This will be examined during: a) an initial four-week treatment with taper; b) a 12-week stabilization treatment for those who do not respond successfully to the initial treatment; and c) a long-term follow-up assessment at 1.5 years, 2.5 years, and 3.5 years after treatment.

DETAILED DESCRIPTION:
This is a randomized 2-phase, open-label; multi-center study conducted in outpatient treatment settings. The main objective of this study is to identify an effective sublingual buprenorphine/naloxone treatment regimen for subjects dependent on prescription opioids. Phase 1 of this study will assess the prevailing one-month detoxification practice. This phase will assess the benefits of individual drug counseling in a short-term treatment paradigm. The second phase of this study will assess the benefit of individual drug counseling in a longer-term treatment paradigm for participants who did not respond successfully to the short-term buprenorphine/naloxone treatment. There is also a long-term follow-up assessment to determine outcomes at 1.5 years, 2.5 years, and 3.5 years after treatment.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older
* Physically dependent on opioids
* Meet DSM-IV criteria for opioid dependence

Exclusion Criteria:

* Known allergy or sensitivity to buprenorphine or naloxone
* Unstable psychiatric disorder
* Pregnant or lactating females
* Liver function test results greater than 5 times the upper limit of normal range

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 653 (Actual)
Dates: Start 2006-05; Primary Completion 2009-07 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roger Weiss, M.D., Principal Investigator — Mclean Hospital; Walter Ling, M.D., Principal Investigator — University of California, Las Angeles
Locations (12):
- United States (12):
  - Integrated Substance Abuse Programs, Los Angeles, California
  - San Francisco General Hospital, San Francisco, California
  - East Indiana Treatment Center, Lawrenceburg, Indiana
  - McLean Hospital, Alcohol and Drug Abuse Treatment Program, Belmont, Massachusetts
  - North Shore - Long Island Jewish Health Systems, Glen Oaks, New York
  - Bellevue Hospital Center, New York, New York
  - St. Luke's Roosevelt Hospital Center, New York, New York
  - ADAPT, Inc., Roseburg, Oregon
  - Behavioral Health Services of Pickens County, Pickens, South Carolina
  - Homeward Bound, Inc., Dallas, Texas
  - Providence Behavioral Health Service, Everett, Washington
  - Chestnut Ridge Hospital, Morgantown, West Virginia

REFERENCES:
- [Background] Weiss RD, Potter JS, Provost SE, Huang Z, Jacobs P, Hasson A, Lindblad R, Connery HS, Prather K, Ling W. A multi-site, two-phase, Prescription Opioid Addiction Treatment Study (POATS): rationale, design, and methodology. Contemp Clin Trials. 2010 Mar;31(2):189-99. doi: 10.1016/j.cct.2010.01.003. Epub 2010 Jan 29. PMID 20116457
- [Background] Potter JS, Prather K, Kropp F, Byrne M, Sullivan CR, Mohamedi N, Copersino ML, Weiss RD. A method to diagnose opioid dependence resulting from heroin versus prescription opioids using the Composite International Diagnostic Interview. Contemp Clin Trials. 2010 Mar;31(2):185-8. doi: 10.1016/j.cct.2010.01.002. Epub 2010 Jan 14. PMID 20079463
- [Background] Weiss RD, Potter JS, Copersino ML, Prather K, Jacobs P, Provost S, Chim D, Selzer J, Ling W. Conducting clinical research with prescription opioid dependence: defining the population. Am J Addict. 2010 Mar-Apr;19(2):141-6. doi: 10.1111/j.1521-0391.2009.00017.x. PMID 20163386
- [Background] Upadhyay J, Maleki N, Potter J, Elman I, Rudrauf D, Knudsen J, Wallin D, Pendse G, McDonald L, Griffin M, Anderson J, Nutile L, Renshaw P, Weiss R, Becerra L, Borsook D. Alterations in brain structure and functional connectivity in prescription opioid-dependent patients. Brain. 2010 Jul;133(Pt 7):2098-114. doi: 10.1093/brain/awq138. Epub 2010 Jun 16. PMID 20558415
- [Background] Dreifuss JA, Griffin ML, Frost K, Fitzmaurice GM, Potter JS, Fiellin DA, Selzer J, Hatch-Maillette M, Sonne SC, Weiss RD. Patient characteristics associated with buprenorphine/naloxone treatment outcome for prescription opioid dependence: Results from a multisite study. Drug Alcohol Depend. 2013 Jul 1;131(1-2):112-8. doi: 10.1016/j.drugalcdep.2012.12.010. Epub 2013 Jan 18. PMID 23333292
- [Result] Weiss RD, Potter JS, Fiellin DA, Byrne M, Connery HS, Dickinson W, Gardin J, Griffin ML, Gourevitch MN, Haller DL, Hasson AL, Huang Z, Jacobs P, Kosinski AS, Lindblad R, McCance-Katz EF, Provost SE, Selzer J, Somoza EC, Sonne SC, Ling W. Adjunctive counseling during brief and extended buprenorphine-naloxone treatment for prescription opioid dependence: a 2-phase randomized controlled trial. Arch Gen Psychiatry. 2011 Dec;68(12):1238-46. doi: 10.1001/archgenpsychiatry.2011.121. Epub 2011 Nov 7. PMID 22065255
- [Derived] McHugh RK, Bailey AJ, McConaghy BA, Weiss RD, Fiellin DA, Hillhouse M, Moore BA, Fitzmaurice GM. Behavioral Therapy as an Adjunct to Buprenorphine Treatment for Opioid Use Disorder: A Secondary Analysis of 4 Randomized Clinical Trials. JAMA Netw Open. 2025 Aug 1;8(8):e2528529. doi: 10.1001/jamanetworkopen.2025.28529. PMID 40833692
- [Derived] Brandt L, Odom GJ, Hu MC, Castro C, Balise RR; CTN-0094 Team. Empirically contrasting urine drug screening-based opioid use disorder treatment outcome definitions. Addiction. 2024 Jul;119(7):1289-1300. doi: 10.1111/add.16494. Epub 2024 Apr 14. PMID 38616571
- [Derived] McDermott KA, Griffin ML, McHugh RK, Fitzmaurice GM, Jamison RN, Provost SE, Weiss RD. Long-term naturalistic follow-up of chronic pain in adults with prescription opioid use disorder. Drug Alcohol Depend. 2019 Dec 1;205:107675. doi: 10.1016/j.drugalcdep.2019.107675. Epub 2019 Oct 28. PMID 31715440
- [Derived] Weiss RD, Griffin ML, Marcovitz DE, Hilton BT, Fitzmaurice GM, McHugh RK, Carroll KM. Correlates of Opioid Abstinence in a 42-Month Posttreatment Naturalistic Follow-Up Study of Prescription Opioid Dependence. J Clin Psychiatry. 2019 Mar 26;80(2):18m12292. doi: 10.4088/JCP.18m12292. PMID 30920187
- [Derived] McDermott KA, Griffin ML, Connery HS, Hilario EY, Fiellin DA, Fitzmaurice GM, Weiss RD. Initial response as a predictor of 12-week buprenorphine-naloxone treatment response in a prescription opioid-dependent population. J Clin Psychiatry. 2015 Feb;76(2):189-94. doi: 10.4088/JCP.14m09096. PMID 25562462
- [Derived] Potter JS, Dreifuss JA, Marino EN, Provost SE, Dodd DR, Rice LS, Fitzmaurice GM, Griffin ML, Weiss RD. The multi-site prescription opioid addiction treatment study: 18-month outcomes. J Subst Abuse Treat. 2015 Jan;48(1):62-9. doi: 10.1016/j.jsat.2014.07.009. Epub 2014 Aug 2. PMID 25189089
- [Derived] Griffin ML, Dodd DR, Potter JS, Rice LS, Dickinson W, Sparenborg S, Weiss RD. Baseline characteristics and treatment outcomes in prescription opioid dependent patients with and without co-occurring psychiatric disorder. Am J Drug Alcohol Abuse. 2014 Mar;40(2):157-62. doi: 10.3109/00952990.2013.842241. Epub 2013 Nov 12. PMID 24219166

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 653 treatment-seeking outpatients dependent on prescription opioids across 10 U.S. sites.
Groups:
- Buprenorphine/Nx With EMM: All study participants received buprenorphine-naloxone. This treatment group (Buprenorphine/Naloxone with Enhanced Medical Management) consisted of Standard Medical Management office visits with study physicians certified to prescribe buprenorphine and opioid drug counseling from a trained substance abuse or mental health professional.
- Buprenorphine/Nx With SMM: All study participants received buprenorphine-naloxone medication. This treatment group (buprenorphine-naloxone with Standard Medical Management) consisted of office visits with study physicians certified to prescribe buprenorphine.
Period: Phase 1 (12 Weeks)
Arm/Group | Buprenorphine/Nx With EMM | Buprenorphine/Nx With SMM
Started | 329 | 324
Completed | 19 | 24
Not Completed | 310 | 300
Not completed — Lost to Follow-up | 88 | 75
Not completed — Investigator-initiated termination | 2 | 0
Not completed — Eligible for Phase 2 | 220 | 225
Period: Phase 2 (24 Weeks)
Arm/Group | Buprenorphine/Nx With EMM | Buprenorphine/Nx With SMM
Started | 180 | 180
Completed | 161 | 161
Not Completed | 19 | 19
Not completed — Lost to Follow-up prior to wk 13 | 19 | 18
Not completed — Discontinued intervention (jailed) | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Buprenorphine/Nx With EMM | Buprenorphine/Nx With SMM | Total
Number analyzed (Participants) | 329 | 324 | 653
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 329 | 324 | 653
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 32.9 (10.1) | 33.5 (10.3) | 33.2 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 125 | 136 | 261
  Male | 204 | 188 | 392
Region of Enrollment [Number; unit: participants]
  United States | 329 | 324 | 653

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants Attaining Successful Opioid Use Outcome by Counseling Condition at End of Phase 1
Description: In Phase 1, successful outcome was defined as completing week 12 with self-reported opioid use on no more than 4 days in a month, absence of 2 consecutive opioid-positive urine test results, no additional substance use disorder treatment (other than self-help), and no more than 1 missing urine sample during the 12 weeks.
Time Frame: 12 weeks
Population: 653 study participants randomized to Phase 1 were included in analysis.
Measure: Number; unit: participants
Arm/Group | Buprenorphine/Nx With EMM | Buprenorphine/Nx With SMM
Number analyzed (Participants) | 329 | 324
participants | 19 [3.5 to 8.9] | 24 [4.8 to 10.8]

2. Secondary Outcome: The Number of Participants Attaining Successful Opioid Use Outcome by Counseling Condition Phase 2, 8-week Posttreatment Follow-up
Description: A planned secondary outcome, successful outcome at week 24, that is, 8 weeks after completion of buprenorphine-naloxone taper, was defined the same as at week 12 of Phase 2, that is abstinent from opioids during week 24 and at least 2 of the previous 3 weeks.
Time Frame: 24 weeks in Phase 2 period (i.e., 36 weeks into the study)
Population: 360 participants randomized to Phase 2 were included in the analysis.
Measure: Number; unit: participants
Arm/Group | Buprenorphine/Nx With EMM | Buprenorphine/Nx With SMM
Number analyzed (Participants) | 180 | 180
participants | 18 | 13

3. Secondary Outcome: The Number of Participants Attaining Successful Opioid Use Outcomes in Phase 1 by Chronic Pain Condition
Description: As a planned secondary analysis, we examined the impact of the two Phase 1 stratification variables on the primary end points. Patients were designated at baseline as having current chronic pain if they reported pain "other than everyday kinds of pain" excluding withdrawal-related pain, for at least 3 months.
Time Frame: 12 weeks
Population: 379 identified as having chronic pain at baseline in Phase 1.
Measure: Number; unit: participants
Groups:
- Success in Phase 1 Among Participants With Chronic Pain: Patients were designated at baseline as having current chronic pain if they reported pain "other than everyday kinds of pain" excluding withdrawal-related pain, for at least 3 months.
Arm/Group | Success in Phase 1 Among Participants With Chronic Pain | Success in Phase 1 Among Participants Without Chronic Pain
Number analyzed (Participants) | 379 | 274
participants | 30 | 13

4. Secondary Outcome: The Number of Participants Attaining Successful Opioid Use Outcomes in Phase 2 by Chronic Pain Condition
Description: as for outcome 3
Time Frame: 12 weeks
Measure: Number; unit: participants
Groups:
- Success in Phase 2 Among Participants With Chronic Pain: Patients were designated at baseline as having current chronic pain if they reported pain "other than everyday kinds of pain" excluding withdrawal-related pain, for at least 3 months.
Arm/Group | Success in Phase 2 Among Participants With Chronic Pain | Success in Phase 2 Among Participants Without Chronic Pain
Number analyzed (Participants) | 149 | 211
participants | 79 | 98

5. Secondary Outcome: The Number of Participants With and Without Any Lifetime Use of Heroin Attaining Successful Opioid Use Outcomes in Phase 1
Description: As a planned secondary analysis, we examined the impact of the two phase 1 stratification variables on the primary outcome.
Time Frame: 12 weeks
Population: Participants randomized to Phase 1 were stratified by two variables: current chronic pain and lifetime heroin use.
Measure: Number; unit: participants
Arm/Group | Success in Phase 1 Among Participants With Heroin Use | Success in Phase 1 Among Participants Without Heroin Use
Number analyzed (Participants) | 150 | 503
participants | 9 | 34

6. Secondary Outcome: The Number of Participants With and Without Any Lifetime Use of Heroin Attaining Successful Opioid Use Outcomes in Phase 2
Description: as for outcome 5
Time Frame: 12 weeks
Measure: Number; unit: participants
Arm/Group | Success in Phase 2 Among Participants With Heroin Use | Success in Phase 2 Among Participants Without Heroin Use
Number analyzed (Participants) | 100 | 260
participants | 37 | 140

7. Primary Outcome: The Number of Participants Attaining Successful Opioid Use Outcome by Counseling Condition, Phase 2 End of Treatment
Description: In phase 2, successful outcome was defined as abstaining from opioids during week 12 (the final week of buprenorphine-naloxone stabilization) and during at least 2 of the previous 3 weeks (weeks 9-11). This outcome measure required substantial improvement but not complete abstinence.
Time Frame: 12 weeks in Phase 2 period (i.e., 24 weeks into the study)
Population: 360 participants randomized to Phase 2 were included in the analysis.
Measure: Number; unit: participants
Arm/Group | Buprenorphine/Nx With EMM | Buprenorphine/Nx With SMM
Number analyzed (Participants) | 180 | 180
participants | 93 | 84

ADVERSE EVENTS:
Time Frame: Adverse Events were captured beginning at the time of randomization and every subsequent research visit.
Arm/Group | Buprenorphine/Nx With EMM | Buprenorphine/Nx With SMM
Serious Adverse Events (participants affected / at risk) | 6/329 | 5/324
Other Adverse Events (participants affected / at risk) | 277/329 | 265/324
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Buprenorphine/Nx With EMM (N=329) | Buprenorphine/Nx With SMM (N=324)
Suicidal Ideation (Psychiatric disorders) | 0 (0) | 2 (2)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Gastric Ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Accidental Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Grand Mal Convulsion (Nervous system disorders) | 1 (1) | 0 (0)
Urinary Retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Ovarian Cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Ovarian Torsion (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Buprenorphine/Nx With EMM (N=329) | Buprenorphine/Nx With SMM (N=324)
Headache (Nervous system disorders) | 108 (130) | 83 (98)
Constipation (Gastrointestinal disorders) | 42 (42) | 62 (64)
Nausea (Gastrointestinal disorders) | 46 (48) | 38 (42)
Insomnia (Psychiatric disorders) | 39 (40) | 47 (48)
Vomiting (Gastrointestinal disorders) | 27 (32) | 30 (32)
Anxiety (Psychiatric disorders) | 30 (30) | 24 (25)
Toothache (Gastrointestinal disorders) | 19 (19) | 22 (25)
Nasopharyngitis (Infections and infestations) | 21 (21) | 15 (17)
Back Pain (Musculoskeletal and connective tissue disorders) | 16 (16) | 24 (26)
Fatigue (General disorders) | 18 (18) | 17 (18)

LIMITATIONS AND CAVEATS:
A treatment providing infrequent or no medical management was not included. It is not known if less intensive medical management would affect outcomes. Length of the trial may have also affected results. Pain severity was only moderate on average.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No